CLINICAL TRIAL: NCT01481064
Title: Effect and Cost Evaluation of a Multifaceted Approach Including Audit and Feedback With a Patient-centredness Questionnaire in Fertility Care.
Brief Title: Effect and Cost Evaluation of a Multifaceted Approach With a Patient-centredness Questionnaire in Fertility Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.G. Huppelschoten (Other)
Responsible Party: Sponsor-Investigator, A.G. Huppelschoten, MD, Principal Investigator, University Medical Center Nijmegen
Organization: University Medical Center Nijmegen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R0000869
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Patient Centredness; Quality of Life; Risk Factors for Emotional Maladjustment
Keywords: Patient centredness; Quality of life; Multifaceted approach; Fertility care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifaceted approach (Active Comparator): After baseline measurement a multifaceted approach will start for 1 year, including audit and feedback, an educational outreach visit, and patient-mediated interventions.
  Interventions: Behavioral: Multifaceted approach
- Usual care (No Intervention): After baseline measurement no intervention will occur in these hospitals.

INTERVENTIONS:
Behavioral: Multifaceted approach — Audit and feedback, educational outreach visits, and patient-mediated interventions.
  Arms: Multifaceted approach

SUMMARY:
The purpose of this study is to evaluate the effects and costs of a multifaceted approach on the patient-centredness of fertility care and the quality of life of fertility patients.

DETAILED DESCRIPTION:
Besides traditional outcomes as (cost)-effectiveness and safety, the Institute of Medicine calls patient-centredness as an independent outcome indicator to evaluate quality of healthcare. Nevertheless, within fertility care there is great variation in the delivery of patient-centred care and room for improvement.

The effects of a multifaceted approach on patient centredness and quality of life will be determined by a baseline and after measurement. Three questionnaires will be used to measure patient centredness (Patient Centredness Questionnaire-Infertility), Quality of Life (FertiQoL) and risk factors of emotional maladjustment(SCREENIVF). The multifaceted approach consists of: 1)audit and feedback, 2) educational outreach visits, and 3) patient-mediated interventions.

During one year the multifaceted approach is performed followed by an after measurement with the same questionnaires. The effects and costs of the multifaceted approach will be determined. Process evaluation will be performed to investigate feasibility and to study wether and to what extend patients and professionals used and appreciated the elements of the multifaceted approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing MAR-treatment (ovulation induction, intra-uterine inseminations, in vitro fertilization, or intra-cytoplasmic sperm injection).

Exclusion Criteria:

* Pregnant couples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the level of patient-centredness at one year | one year
  Main outcome measure will be the difference in the level of patient-centredness after the multifaceted approach between control and intervention group. The level of patient-centredness will be determined by a patients' questionnaire (PCQ-Infertility).

SECONDARY OUTCOMES:
Change from baseline in patients' quality of life at one year | 1 year
  Differences in the level of quality of life at after measurement between control and intervention group will be determined.
Change from baseline in risk factors of emotional maladjustment at one year | 1 year
  Differences in risk factors of emotional maladjustment at after measurement between control and intervention group will be determined.
Cost-effectiveness | one year
  A cost-effectiveness analysis will be performed to evaluate efficiency of the multifaceted approach at different thresholds (cost-effectiveness acceptibility curve)

CONTACTS AND LOCATIONS:
Overall Officials: J Kremer, PhD, Study Chair — Radboud University Medical Center; W Nelen, PhD, Study Director — Radboud University Medical Center; A Huppelschoten, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Radboud Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Huppelschoten AG, Nelen WL, Westert GP, van Golde RJ, Adang EM, Kremer JA. Improving patient-centredness in partnership with female patients: a cluster RCT in fertility care. Hum Reprod. 2015 May;30(5):1137-45. doi: 10.1093/humrep/dev041. Epub 2015 Mar 6. PMID 25750102
- [Derived] Huppelschoten AG, van Duijnhoven NT, Hermens RP, Verhaak C, Kremer JA, Nelen WL. Improving patient-centeredness of fertility care using a multifaceted approach: study protocol for a randomized controlled trial. Trials. 2012 Sep 24;13:175. doi: 10.1186/1745-6215-13-175. PMID 23006997